CLINICAL TRIAL: NCT03893357
Title: Retrospective Study of the Prevalence of Antiphospholipid Antibodies in the Population of Hemodialysis Patients at the CHU Brugmann Hospital
Brief Title: Prevalence of Antiphospholipid Antibodies in the Hemodialysis Patients Population Within the CHU Brugmann Hospital
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Agnieszka Pozdzik, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Fatim
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for antiphospholipid antibodies: Patients tested positive for antiphospholipid antibodies
  Interventions: Other: Data extraction from medical files
- Negative for antiphospholipid antibodies: Patients tested negative for antiphospholipid antibodies
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Retrospective data extraction from the medical files

SUMMARY:
In patients with a chronic renal disease at the terminal stage, extrarenal epuration is essential for the control of clinico-biological complications. Two extrarenal epuration techniques are currently available: peritoneal dialysis (using the peritoneal membrane of the patient) and hemodialysis, requiring the use of an external biocompatible membrane known as 'dialysis filter'. This technique requires a vascular access (arteriovenous fistula or dialysis catheter). The thrombosis of vascular accesses represents a major cause of morbidity and mortality in hemodialysis patients. Thrombosis are more frequent when using synthetic prosthetic arteriovenous fistula instead of native arteriovenous fistula.

Antiphospholipid Syndrome (APLS) is a rare autoimmune disease characterized by arterial thrombosis, venous thrombosis and obstetrical complications such as as defined by the Sidney's criteria.

In the general population, the presence of antiphospholipid antibodies is associated with an increased risk of thromboembolic events. In the nephrological population, this prevalence is higher in hemodialysis patients compared to patients on peritoneal dialysis or non-dialyzed patients. Up to 37% of hemodialysis patients are positive for antiphospholipid antibodies and this biology is associated with thrombotic events and vascular access thromboses. However, some studies do not report this association and there is currently no consensus in terms of the therapeutic management of these patients.

Some factors influencing the positivity for antiphospholipid antibodies have been reported: smoking, age, the presence of a non-glomerular nephropathy, hypoalbuminaemia, the use of a central venous catheter for dialysis or the use of a non-biocompatible dialysis membrane.

Taking into account the conflicting data from the literature, it seems important to study the respective role(s) of 3 types of antiphospholipid antibodies in the occurrence of thrombo- embolic events in patients undergoing dialysis within the CHU Brugmann Hospital.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing dialysis within the CHU Brugmann Hospital

Exclusion Criteria:

* Mutation of factor V
* Mutation G20210A of the prothrombin gene
* Protein C deficiency
* Protein S deficiency
* Antithrombin III deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing dialysis within the CHU Brugmann Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of antiphospholipid antibodies | 19 years
  Prevalence of antiphospholipid antibodies
Prevalence of arterial thrombosis | 19 years
  Prevalence of arterial thrombosis
Prevalence of venous thrombosis | 19 years
  Prevalence of venous thrombosis
Maturation delay of the arteriovenous fistula | 19 years
  Maturation delay of the arteriovenous fistula
Percentage of thrombosis of the filter | 19 years
  Percentage of thrombosis of the filter
Lifespan of the catheter | 19 years
  Lifespan of the catheter
Lifespan of the fistula | 19 years
  Lifespan of the fistula

SECONDARY OUTCOMES:
Existence of thrombosis risk factors | 19 years
  Existence of at least one of the following pro-thrombotic risk factors: smoking, active neoplasia, arterial hypertension.
Anticoagulant treatment | 19 years
  Existence of an anticoagulant treatment
  Presence of an anticoagulant treatment by means of anti-vitamin K
Antiplatelet treatment Antiplatelet treatment | 19 years
  Existence of an antiplatelet treatment
Antihypertensive treatment | 19 years
  Existence of an antihypertensive treatment
Statin treatment | 19 years
  Existence of a treatment by means of statins
Ethiology of the nephropathy (known/unknown) | 19 years
  Known versus unknown ethiology
Ethiology of the nephropathy (glomerular) | 19 years
  Glomerular versus non-glomerular ethiology
Age at dialysis entry | 19 years
  Age at dialysis entry
Vascular access | 19 years
  Catheter versus distal arteriovenous fistula versus proximal arteriovenous fistula
Type of dialysis | 19 years
  Hemodiafiltration versus conventional hemodialysis
Type of per-dialytic anticoagulation | 19 years
  With or without heparin
Brand of dialysis membrane | 19 years
  Brand of dialysis membrane
Urea change percentage | Last available result within 19 years
  Urea change percentage
Activated partial thromboplastin time (aPTT) | Last available result within 19 years
  Coagulation assessment
Hemoglobin count | Last available result within 19 years
  Hemoglobin count
Platelets count | Last available result within 19 years
  Platelets count

CONTACTS AND LOCATIONS:
Overall Officials: Camara Fatim, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No